CLINICAL TRIAL: NCT01404338
Title: An Investigator-Initiated, Double-Blind, Vehicle-Controlled Study: Assessment for Tachyphylaxis to Topical Corticosteroids in the Treatment of Psoriasis
Brief Title: Assessment for Tachyphylaxis to Topical Corticosteroids in the Treatment of Psoriasis
Acronym: Tachyphylaxis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Patel, Rita Vikram, M.D. (Individual)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Basic Science
Other Study IDs: 11-0422
Record Dates: First submitted 2011-07-25; First posted 2011-07-28 (Estimated); Last update posted 2011-07-28 (Estimated); Status verified 2011-07

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — halobetasol; Ointments

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active Arm (Active Comparator): 1. Active arm/Target Lesion: Halobetasol 0.05% ointment applied under occlusion to be left in place for one week
  Interventions: Drug: Halobetasol 0.05% ointment
- Vehicle Arm (Placebo Comparator): Vehicle arm/Comparator Lesion: Vehicle ointment applied under occlusion to be left in place for one week
  Interventions: Drug: Placebo Ointment

INTERVENTIONS:
Drug: Halobetasol 0.05% ointment
  Arms: Active Arm
Drug: Placebo Ointment
  Arms: Vehicle Arm

SUMMARY:
Tachyphylaxis occurs when a medication is applied multiple times and a decreased response takes place. Many dermatologists believe that tachyphylaxis to topical steroids commonly occur. Other believe that tachyphylaxis can be explain by patient non-compliance with topical medications. This study is looking to prove or disprove the phenomenon of tachyphylaxis by using topical steroids in the psoriasis patient population. The investigators are looking to enroll 10 patients with symmetric, bilateral, and small psoriasis plaques. The investigators will either apply a strong topical steroid or a vehicle ointment to the plaques, which is be occluded with a band aid for a one week period. Weekly, the investigators will inspect the plaques for tachyphylaxis. This regimen will be repeated during phase 2, to see if there is change in the time to tachyphylaxis. This regimen will be repeated during phase 3, however, both plaques will be treated with steroid in this phase, and time to tachyphylaxis will be measured.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be at least 18 years of age and in good general health as confirmed by a medical history.
* Females of childbearing potential must have a negative urine pregnancy test on Baseline/Week 0 and must agree to use adequate birth control methods during the entire study (a barrier method i.e. condoms, diaphragm; hormonal contraceptives i.e. birth control pills, implants, or injections; intrauterine device, or abstinence).
* Subjects must be diagnosed with stable plaque psoriasis affecting 1% to 10% body surface area (excluding the face, scalp, groin, axillae or other intertriginous areas).
* Subjects receiving phototherapy for their psoriasis.
* Subjects must have at least two symmetrical lesions suitable for evaluating response to test agents (one on the right side and one on the left side of the body). The severity of the disease for each target lesion at Baseline/Week 0 must be rated at least 2 (Mild) for each of the key psoriasis characteristics (scaling, erythema, and plaque elevation) on the Target Lesion Severity Score.
* Subjects must be able to understand the requirements of the study abide by the restrictions and return for the required examinations.

Exclusion Criteria:

* Female subjects who are pregnant, nursing or planning a pregnancy during the study.
* Subjects with known hypersensitivity to any components of the test medication.
* Subjects with non-plaque psoriasis (e.g. guttate, erythrodermic) or other related diseases not classified as plaque psoriasis.
* Subjects whose psoriasis involves only the scalp, face, groin, axillae, and/or other intertriginous areas.
* Subjects requiring any other medication (topical or systemic) that may affect the course of the disease during the study period as determined by the study investigators.
* Subjects using biologics or any other systemic treatment (e.g. immunosuppressants, acitretin) for psoriasis within 12 weeks of entering the study.
* Subjects using systemic corticosteroids within 28 days of entering the study
* Subjects using topical corticosteroids or other topical therapies (other than emollients) at the treatment area locations within 14 days of entering the study
* Subjects using phototherapy (UVB, PUVA) on target treatment sites within 4 weeks of entering the study.
* Subjects with overt pre-existing telangiectasias or skin atrophy at intended treatment sites (treatment areas).
* Subjects who are using any medication or has any disease which in the judgment of the investigator will interfere with the conduct or interpretation of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2011-06

PRIMARY OUTCOMES:
Time to Tachyphylaxis | 4 Weeks
  Phase 1: %change in TLSS of target lesion versus comparator lesion Phase 2a, after an interim discontinuation period of 4-8 weeks: %change in TLSS of target lesion versus comparator lesion Phase 2b, after an interim discontinuation period of 4-8 weeks: Percent change in TLSS of the comparator lesion (now switched to open-label halobetasol 0.05% ointment) versus target lesion